CLINICAL TRIAL: NCT06557187
Title: Hippocampus-Avoidance Whole-Brain Radiation Therapy With Simultaneous Integrated Boost for Multiple Brain Metastases in Non-small Cell Lung Cancer
Brief Title: Hippocampus-Avoidance Whole-Brain Radiation Therapy With Simultaneous Integrated Boost for BMs of NSCLC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yatian Liu (Other)
Responsible Party: Sponsor-Investigator, Yatian Liu, Associate Professor in Nanjing Medical University and Deputy chief physician in Jiangsu Cancer Hospital, Jiangsu Cancer Institute & Hospital
Organization: Jiangsu Cancer Institute & Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JZ233490202001088; 100000RMB (Other Grant/Funding Number: Nanjing Medical University of Collaborative Center)
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Brain Metastases; Non-small Cell Lung Cancer
Keywords: brain metastases; hippocampus-avoidance; whole-brain radiation therapy; simultaneous integrated boost
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hippocampus-Avoidance Whole-Brain Radiation Therapy With Simultaneous Integrated Boost (Experimental): HA-WBRT (30 Gy in 12 fractions, Dmax of the hippocampal volume ≤ 17 Gy, Dmean of the hippocampal volume ≤12 Gy) +SIB (48 Gy in 12 fractions)
  Interventions: Radiation: ippocampus-Avoidance Whole-Brain Radiation Therapy With Simultaneous Integrated Boost

INTERVENTIONS:
Radiation: ippocampus-Avoidance Whole-Brain Radiation Therapy With Simultaneous Integrated Boost — hippocampus-Avoidance Whole-Brain Radiation Therapy With Simultaneous Integrated Boost

SUMMARY:
WBRT (whole-brain radiation therapy) exhibits poor tumor control and decreased NCF (neurocognitive function). Herein, we investigated the safety and efficacy of HA-WBRT+SIB (hippocampus-avoidance whole-brain radiation therapy with simultaneous integrated boost) in NSCLC (non-small cell lung cancer) with multiple brain metastases.We conducted a prospective, single-arm phase II trial administering HA-WBRT (30 Gy in 12 fractions, Dmax of the hippocampal volume ≤ 17 Gy, Dmean of the hippocampal volume ≤12 Gy) +SIB (48 Gy in 12 fractions) for multiple brain metastases (≥4) of NSCLC. Cognitive performance was assessed by the HVLT-R DR (Hopkins Verbal LearningTest-Revised delayed Recall).A-WBRT+SIB emerges as a promising and safe therapeutic, improving intracranial tumor control and protecting cognitive function in NSCLC with multiple brain metastases.

DETAILED DESCRIPTION:
Lung cancer has high incidence and mortality rates. NSCLC is the most prevalent form accounting for 85% of all lung cancer cases with approximately 40% of individuals developing brain metastases during the illness. With advancements in therapies like targeted therapy and immunotherapy, the incidence of brain metastases have raised paralleled by a rise in survival rates of NSCLC. And NSCLC patients with brain metastases only 2 to 3 months of natural survival[6]. Therefore, it is urgent to improve the prognosis and intracranial control of NSCLC patients with brain metastases.

Brain metastases patients of NSCLC should be treated with local treatment on the basis of systemic treatment. For patients of NSCLC with brain metastases who are not suitable for targeted therapy or with progressing intracranial post targeted therapy, radiotherapy emerges as a significant therapeutic.Stereotactic radiosurgery (SRS) alone should be offered to patients with one to three unresected brain metastases for patients with asymptomatic brain metastases and no systemic therapy options.While the standard treatment for multiple brain metastases (≥4) remains controversial.

WBRT is used to be a common therapy in multiple brain metastases prolonging survival of patients to 6 months. But WBRT comes with neurotoxic effects, notably cognitive impairment affecting memory and learning. This cognitive decline is mainly attributed to hippocampal damage, a crucial region for learning and memory. The RTOG0933 and NRG Oncology CC001 trials have demonstrated that HA-WBRT effectively safeguards cognitive function and enhances the quality of life in patients with brain metastases. Furthermore, considering the tolerated dose of normal brain tissue, the dose of WBRT was low (30Gy/10F) with only 60% intracranial local control rate. The landmark RTOG9508 trial has demonstrated that WBRT in combination with boosted metastases can improve local intracranial control.

Prokic et al. reported that the simultaneous integrated boost during WBRT (WBRT+SIB) demonstrated superior hippocampal sparing and biological benefits of fractionation over sequential integrated boost. Advancements in radiotherapy techniqueshave led to the innovative HA-WBRT+SIB strategy, delivering higher dosages to existing metastases while minimizing radiation exposure to the hippocampus. However, evidence for the application of HA-WBRT+SIB in multiple (≥4) brain metastases of NSCLC remains insufficient. Therefore, this study aims to investigate the efficacy and safety of HA-WBRT+SIB in patients with multiple brain metastases of NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* adults (aged 18-75 years) diagnosed with NSCLC, with a KPS (Karnofsky performance status) ≥70, at least four brain metastases visible on MRI (magnetic resonance imaging) outside a 5-mm margin around the bilateral hippocampi, not suitable for targeted therapy or progressing intracranial post targeted therapy.

Exclusion Criteria:

* Ineligible participants had a history of conditions affecting cognitive function (including mental illness, brain trauma, and Alzheimer's disease), other primary malignant tumors, uncontrolled systemic disease, uncontrolled extracranial sites of gross disease, and suitable for targeted therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial local progression-free survival time (iLPFS) | From date of enrollment until the date of progression of existing intracranial metastases or date of death from any cause, whichever came first, assessed up to 20 months
  determined as the time from HA-WBRT+SIB initiation to death, existing intracranial metastases progression, or last follow-up.

SECONDARY OUTCOMES:
Intracranial progression-free survival time (iPFS) | From date of enrollment until the date of progression of existing or new metastases intracranial or date of death from any cause, whichever came first, assessed up to 20 months
  measured from HA-WBRT+SIB initiation to existing or new metastases intracranial progression, death, or last follow-up.
Cognitive function | From enrollment to the end of treatment at 4 weeks
  was measured by the relative change in HVLT-R DR score from the start of HA-WBRT+SIB to 4 months after the start of HA-WBRT+SIB.
OS (Overall survival) | From date of enrollment until the date of death from any cause, whichever came first, assessed up to 20 months
  described as the time from initiation of radiation to the last follow-up or death
The cumulative incidence of local intracranial failure | From date of enrollment until the date of progression of existing intracranial metastases， assessed up to 20 months
  measured as the progression of existing intracranial metastases
Cumulative incidence of intracranial failure | From date of enrollment until the date of the progression of existing or new intracerebral metastases assessed up to 20 months
  described as the progression of existing or new intracerebral metastases.

CONTACTS AND LOCATIONS:
Locations (1):
- Yatian Liu, Nanjing, China

IPD SHARING:
Plan to Share IPD: No
The results of the study have not been published